CLINICAL TRIAL: NCT06411223
Title: Project Tara: Pharmacist-led Intervention for Injectable HIV Treatment for Women With Health-related Social Needs
Brief Title: Pharmacist-led Intervention for Injectable HIV Treatment for Women With Health-related Social Needs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000036673
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hiv
Keywords: Criminal legal involvement; Unstably housed; unhoused; Food insecurity; Mental health; Substance use/ treatment engagement; women; Long-acting injectable antiretroviral treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Well-Being | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Intervention Model Description: This is a single-arm prospective interventional pilot study. This study uses a hybrid type 3 implementation study design to evaluate an enhanced pharmacist-led collaborative drug therapy management model (CDTM+) for women with health-related social needs (HRSN), in terms of implementation (primary) and clinical (secondary) outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacist lead CDTM+ (Other): Participants will meet with a clinic-based pharmacist via telehealth for an introductory visit to discuss CAB/RPV LA and possible switch from oral to injectable therapy. The tele-visit can occur by phone or video visit.
  Interventions: Behavioral: Collaborative drug therapy management model; Drug: Cabotegravir/Rilpivirine

INTERVENTIONS:
Behavioral: Collaborative drug therapy management model — CDTM+ is an interdisciplinary approach to patient care in which clinicians collaborate with pharmacists to provide and manage patient drug therapy.
  Other Names: CDTM+
Drug: Cabotegravir/Rilpivirine — Long-acting injectable treatment prescribed to treat HIV-1 infection in people 12 years and older and who weigh at least 77 lbs (35kg), to replace their current HIV-1 medicines when their healthcare provider determines they meet certain requirements.
  Other Names: CAB/RPV LA

SUMMARY:
This study addresses real-world use of long-acting injectable cabotegravir/rilpivirine (CAB/RPV LA) by evaluating implementation and clinical outcomes of a pharmacist-led collaborative drug therapy management model (CDTM+) that will be expanded for telehealth outreach to women with health-related social needs (HRSN).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the implementation and delivery of CAB/RPV LA to women with HRSN by adopting a pharmacist-led CDTM. The project primarily addresses the real-world use of CAB + RPV LA among women who are under-represented in clinical trials and assesses the feasibility and acceptability of CDTM+, and adoption of CAB/RPV LA among participants receiving the CDTM+ model.

Investigators will enhance the existing CDTM to reduce important social and structural barriers to CAB/RPV LA for women with HRSN, by increasing accessibility- using telehealth to deliver CDTM outreach to clinical and community sites without a clinician referral (CDTM+), which is highly scalable. In addition to assessing engagement with the CDTM+ intervention and impact on key implementation (reach, feasibility, acceptability, uptake) and clinical outcomes (CAB/RPV LA initiation), investigators will also assess impact on patient engagement in non-HIV related care and psychological, sexual, and social well-being.

ELIGIBILITY:
Inclusion Criteria:

* Living with diagnosed HIV
* Receiving HIV care-related services from Yale New Haven Health (YNHH)
* Currently on oral ART and virally suppressed for at least 6 months (from electronic health review).
* Have experienced at least one HRSN: a) homelessness or housing insecurity; b) food insecurity; c) criminal legal system involvement; OR d) substance use in the past 3 years (from self-report at screening).
* Able to converse comfortably in English or Spanish

Exclusion Criteria:

* Unable or unwilling to complete informed consent (e.g., have a conservator of person)
* Have initiated CAB/RPV oral lead-in prior to enrollment.
* Have a contraindication to CAB/RPV LA per label.
* Have known or suspected resistance to CAB/RPV
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female (cis- or trans-)
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of CDTM+ | Baseline, Month 12
  Feasibility of CDTM+ assessed using the Intervention Measure: 4-item Likert scale, each item scored 1 (completely disagree) to 5 (completely agree) and averaged. Score range 4-20, higher scores reflect higher feasibility.
Acceptability of CDTM+ | Baseline, Month 12
  Assessed using the Theoretical Framework of Acceptability Questionnaire: 7-items, each scored on Likert scale 1 to 5 and averaged. Score range 7-35, higher scores reflect higher acceptability.
Evaluate the adoption of CAB/RPV LA in the population receiving CDTM+ | Month 12
  Assessed by the percentage of patients who have a documented 1st injection visit

SECONDARY OUTCOMES:
Evaluate the effectiveness of the CDTM+ intervention on intention to switch to CAB/RPV LA | Baseline, immediately following CDTM+
  How likely are you to switch from your current medication to CAB/RPV LA? 5-item Likert scale (1=not at all likely to 5=very likely; score range 1-5)
Among those who initiate CAB/RPV LA, evaluate the effectiveness of CDTM+ on CAB/RPV LA adherence | Month 12
  Percent of on-time injections
Among those who initiate CAB/RPV LA, evaluate the effectiveness of CDTM+ on CAB/RPV LA maintenance of virologic suppression | Month 12
  Percent of participants with HIV VL <50
Reach/penetration of the CDTM+ intervention | Baseline, Month 12
  Enrollment rate (# of people enrolled/# of people screened for eligibility)
Uptake/adoption of the CDTM+ intervention | Baseline, Month 12
  Interaction time*frequency
Barriers and facilitators to CAB/RPV LA initiation | Baseline, Month 6, Month 12
  Qualitative patient interview will be conducted to assess Barriers and facilitators to CAB/RPV LA initiation

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Meyer, MD, MS, FACP, Principal Investigator — Yale University
Locations (1):
- Yale Clinical and Community Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loeliger KB, Altice FL, Desai MM, Ciarleglio MM, Gallagher C, Meyer JP. Predictors of linkage to HIV care and viral suppression after release from jails and prisons: a retrospective cohort study. Lancet HIV. 2018 Feb;5(2):e96-e106. doi: 10.1016/S2352-3018(17)30209-6. Epub 2017 Nov 27. PMID 29191440
- [Background] Philbin MM, Bergen S, Parish C, Kerrigan D, Kinnard EN, Reed S, Cohen MH, Sosanya O, Sheth AN, Adimora AA, Cocohoba J, Goparaju L, Golub ET, Vaughn M, Gutierrez JI Jr, Fischl MA, Alcaide M, Metsch LR. Long-Acting Injectable ART and PrEP Among Women in Six Cities Across the United States: A Qualitative Analysis of Who Would Benefit the Most. AIDS Behav. 2022 Apr;26(4):1260-1269. doi: 10.1007/s10461-021-03483-7. Epub 2021 Oct 14. PMID 34648131
- [Background] Messer LC, Quinlivan EB, Parnell H, Roytburd K, Adimora AA, Bowditch N, DeSousa N. Barriers and facilitators to testing, treatment entry, and engagement in care by HIV-positive women of color. AIDS Patient Care STDS. 2013 Jul;27(7):398-407. doi: 10.1089/apc.2012.0435. PMID 23829330
- [Background] Orkin C, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Overton ET, Girard PM, Oka S, Walmsley S, Bettacchi C, Brinson C, Philibert P, Lombaard J, St Clair M, Crauwels H, Ford SL, Patel P, Chounta V, D'Amico R, Vanveggel S, Dorey D, Cutrell A, Griffith S, Margolis DA, Williams PE, Parys W, Smith KY, Spreen WR. Long-Acting Cabotegravir and Rilpivirine after Oral Induction for HIV-1 Infection. N Engl J Med. 2020 Mar 19;382(12):1124-1135. doi: 10.1056/NEJMoa1909512. Epub 2020 Mar 4. PMID 32130806
- [Background] Swindells S, Andrade-Villanueva JF, Richmond GJ, Rizzardini G, Baumgarten A, Masia M, Latiff G, Pokrovsky V, Bredeek F, Smith G, Cahn P, Kim YS, Ford SL, Talarico CL, Patel P, Chounta V, Crauwels H, Parys W, Vanveggel S, Mrus J, Huang J, Harrington CM, Hudson KJ, Margolis DA, Smith KY, Williams PE, Spreen WR. Long-Acting Cabotegravir and Rilpivirine for Maintenance of HIV-1 Suppression. N Engl J Med. 2020 Mar 19;382(12):1112-1123. doi: 10.1056/NEJMoa1904398. Epub 2020 Mar 4. PMID 32130809
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Meyer JP, Price CR, Ye Y, Qin Y, Tracey D, Demidont AC, Melbourne K, Altice FL. A PrEP Demonstration Project Using eHealth and Community Outreach to Justice-Involved Cisgender Women and Their Risk Networks. AIDS Behav. 2022 Dec;26(12):3807-3817. doi: 10.1007/s10461-022-03709-2. Epub 2022 Jun 7. PMID 35672552
- [Background] Baker O, Wellington C, Price CR, Tracey D, Powell L, Loffredo S, Moscariello S, Meyer JP. Experience delivering an integrated service model to people with criminal justice system involvement and housing insecurity. BMC Public Health. 2023 Feb 2;23(1):222. doi: 10.1186/s12889-023-15108-w. PMID 36732685
- [Background] Harsono D, Deng Y, Chung S, Barakat LA, Friedland G, Meyer JP, Porter E, Villanueva M, Wolf MS, Yager JE, Edelman EJ. Correction to: Experiences with Telemedicine for HIV Care During the COVID-19 Pandemic: A Mixed-Methods Study. AIDS Behav. 2023 Jun;27(6):2054. doi: 10.1007/s10461-022-03907-y. No abstract available. PMID 36318433